CLINICAL TRIAL: NCT01307072
Title: Compliance to Ophthalmic Follow-up Examinations Affect Outcome of Vitrectomy for Proliferative Diabetic Retinopathy
Brief Title: Compliance to Ophthalmic Follow-up Examinations and Surgical Outcome for Proliferative Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Other Study IDs: Kyorineye003
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: periodic examinations, compliance
MeSH Terms: conditions — Patient Compliance | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Never-treated group: The patients who had no previous ophthalmic examination until the first visit when vitreous surgery was prescribed
  Interventions: Procedure: Vitrectomy
- The non-compliant group: The patients with a history of missing ophthalmic examination over a one year period
  Interventions: Procedure: Vitrectomy
- The compliant group: The patients who had ophthalmic examinations at least once a year
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy — Vitrectomy. Diabetic retinopathy
  Other Names: Compliance of follow-up

SUMMARY:
The relationship between the surgical outcome of vitreous surgery for proliferative diabetic retinopathy and the compliance to ophthalmic follow-up examinations was evaluated.

DETAILED DESCRIPTION:
The medical records of 94 patients that had undergone vitreous surgery for proliferative diabetic retinopathy (PDR) and were followed for at least 6 months were reviewed. The subjects were divided into three groups; the never-treated group consisting of patients who had no previous ophthalmic examination until the first visit when vitreous surgery was prescribed; the non-compliant group consisting of patients with a history of missing ophthalmic examination over a one year period, and the compliant group consisting of patients who had ophthalmic examinations at least once a year. The evaluations included age, gender, plasma level of glycosylated hemoglobin (HbA1c) at the preoperative examination, presence of preoperative panretinal photocoagulation, preoperative best-corrected visual acuity (BCVA), postoperative BCVA at the final examination, status of the PDR, the numbers of vitreous surgeries, and presence of pre- and postoperative neovascular glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* One hundred and twenty-eight eyes of 94 patients that had undergone vitreous surgery for proliferative diabetic retinopathy.
* Type 2 diabetes.

Exclusion Criteria:

* The patients were not followed more than 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients that underwent their first vitreous surgery for proliferaftive diabetic retinopathy
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Preoperative status | Preoperative period
  Plasma level of glycosylated hemoglobin (HbA1c)
Preoperative status | Preoperative period
  Best-corrected visual acuity (BCVA),

SECONDARY OUTCOMES:
Postoperative status | up to 1 year
  Postoperative best-corrected visual acuity (BCVA) at 6 months and the final examination
Postoperative status | up to 1 year
  Status of the proliferative diabetic retinopathy
Postoperative status | up to 1 year
  Presence of neovascular glaucoma.

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan